CLINICAL TRIAL: NCT02389907
Title: Assessing the Association Between Patients' Perceptions of Success With Post-Operative Pain Management and Overall Experience With Care
Brief Title: Association Between Patients' Perceptions of Success in Post-op Pain Management and Overall Experience With Care
Status: Withdrawn | Type: Observational
Why Stopped: The study was not developed due to the cessation of IONSYS marketing
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDCO-ERA-14-01
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Total Hip Replacement Group: Adults who have undergone a total hip replacement
- Hysterectomy Group: Adults who have undergone a hysterectomy

SUMMARY:
Assessing the association between patients' perceptions of success with post-operative pain management and overall experience with care.

DETAILED DESCRIPTION:
A study to assess the association between patients' perceptions of success with post-operative pain management following total hip replacement or hysterectomy surgery and their later perception of pain management while in the hospital and the hospital overall.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Subject (or their legally acceptable representative) must have signed an informed consent form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Subject is receiving a unilateral total hip replacement or a hysterectomy (total abdominal hysterectomy, total abdominal hysterectomy/bilateral salpingo-oophorectomy, total vaginal hysterectomy, or total vaginal hysterectomy/salpingo-oophorectomy)
* Subject is expected to remain hospitalized for at least 24 hours post-operatively
* Subject is expected to experience pain requiring IV PCA or non-PCA (non-patient controlled opioids via IV, IM, SC, or PO routes of administration) opioids for at least 24 hours after surgery
* Subject is classified as American Society of Anesthesiology (ASA) category I, II, or III
* Subject is willing to complete the required post-operative survey measures to be completed in the hospital
* Subject is willing to complete a post-discharge survey (including HCAHPS survey instrument) via telephone approximately two-weeks (14 days) post-discharge

Exclusion Criteria:

* Subject is having an operation other than the surgical procedures selected for inclusion (e.g., bilateral or partial hip replacement, or hip revision)
* Subject cannot read, write, and communicate in English
* Subject has a history of tolerance to opioids including those prescribed opioids in the 3 month period leading up to the perioperative period (i.e., a subject is considered to have a potential tolerance to opioids if for 4 consecutive days prior to surgery they have been taking a short acting/short acting combination opioid analgesic greater than 120 mg codein daily, 40 mg hydrocodone daily, 200 mg tramadol daily, or 40 mg oxycodone daily or if they were on any dose of strong opioid analgesic such as morphine, hydromorphone, or fentanyl)
* Subject has a history of allergy to opioids reported pre-operatively or documented in medical history
* Subject is scheduled to receive additional surgical procedures beyond those listed within 72 hours of the initial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include adults 18 years of age or older who have undergone either a total hip replacement or hysterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Patient Global Assessment (PGA) and Hospital Consumer Assessment of Healthcare providers and Systems (HCAHPS) | 24 hours - 14 days post discharge
  Assess the association between patients' perceptions of success with opioid post-operative pain management following total hip replacement or hysterectomy surgery as measured by a patient global assessment (PGA) at 24 hours post-op and at 48 hours post-op, and their perception of pain management while in the hospital and the hospital overall, as measured by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) instrument two-weeks (14 days) post-discharge

SECONDARY OUTCOMES:
Post-Operative Pain Management Modality | 14 days post discharge
  Determine whether there are differences in patients' perception of pain management while in the hospital and the hospital overall with respect to post-operative pain management modality

OTHER OUTCOMES:
Composite outcome measures consisting of multiple measures | 48 Hours Post Op
  Depending on available statistical power, other relevant constructs, including pain severity and mobility, as measured by BPI, a one-item Pain Numerical Rating Scale (NRS), and mobility items from the Ease of Care (EOC) Questionnaire, as well as patient demographic characteristics and medical/medication history will be taken into account when assessing the primary and secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Abraham, MSPT, MBA, Study Director — The Medicines Company
Locations (9):
- United States (9):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Jupiter Medical Center, Jupiter, Florida
  - Phoenix Clinical Research LLC, Tamarac, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Drexel University, Philadelphia, Pennsylvania
  - Magee-Women's Hospital (UPMC), Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Health Research Institute, Fort Worth, Texas

REFERENCES:
- [Result] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Result] Cohen, J. (1988). Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ: Lawrence Earlbaum Associates.